CLINICAL TRIAL: NCT06777836
Title: The Effects of Discharge Education on Patient Satisfaction and Diabetes Empowerment in Diabetic Surgical Patients
Brief Title: Discharge Education in Diabetic Surgical Patients
Acronym: DEDES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ganime Esra Soysal, Assistant Professor, Surgical Nursing, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SBF-HMS-GES-05
Record Dates: First submitted 2025-01-04; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: To Examine the Effects of Diabetes-based Personalised Discharge Education Given to Diabetic Surgical Patients on Satisfaction; To Examine the Effects of Diabetes-based Personalised Discharge Education Given to Diabetic Surgical Patients on Diabetes Empowerment
Keywords: diabetes empowerment; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This study utilizes a randomized experimental design to investigate the effects of discharge education on patient satisfaction and diabetes empowerment among diabetic surgical patients. A sample size of 110 patients will be included, accounting for potential dropouts. Patients will be randomly assigned to receive Personalised Discharge training focused on diabetes management, including blood glucose control, diet, exercise, and medication management. The intervention's outcomes will be measured using validated tools, such as the Discharge Training Satisfaction Scale and the Diabetes Empowerment Scale. Statistical analysis will be conducted using SPSS software to evaluate the efficacy of the intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardised discharge training (No Intervention): Discharge training will be given according to the standard operation.
  Scales to be applied:
  Discharge Training Satisfaction Scale for Surgical Patients: It is a scale developed to measure the satisfaction of surgical patients with discharge training. It consists of 21 items in a five-point Likert structure and has been evaluated as a valid and reliable tool for measuring patient satisfaction. The scale covers factors such as discharge process, personal information, home care, infection monitoring and controls. Cronbach's α reliability coefficient was found to be 0.91, indicating that the scale is highly reliable Diabetes Empowerment Scale: It is a 5-point Likert-type scale consisting of 8 items. Turkish validity and reliability was carried out in 2020 by Jahanpeyma et al.
- Personalised Discharge training (Experimental): In addition to the discharge training given according to the standard surgery, Personalised Discharge training will be given with a holistic patient perspective for diabetes.
  Scales to be applied:
  Discharge Training Satisfaction Scale for Surgical Patients: It is a scale developed to measure the satisfaction of surgical patients with discharge training. It consists of 21 items in a five-point Likert structure and has been evaluated as a valid and reliable tool for measuring patient satisfaction. The scale covers factors such as discharge process, personal information, home care, infection monitoring and controls. Cronbach's α reliability coefficient was found to be 0.91, indicating that the scale is highly reliable Diabetes Empowerment Scale: It is a 5-point Likert-type scale consisting of 8 items. Turkish validity and reliability was carried out in 2020 by Jahanpeyma et al.
  Interventions: Device: Personalised Discharge training

INTERVENTIONS:
Device: Personalised Discharge training — Discharge education also contributes to the empowerment of diabetic surgery patients in diabetes management. During the training process, patients will be informed about blood glucose control, diet, exercise and medication management.
  Arms: Personalised Discharge training

SUMMARY:
In the literature, it is seen that the discharge education given to patients with diabetes is especially focused on the effects of blood glucose control and self-efficacy, and there is no study examining the effects of discharge education on diabetes empowerment with a more general perspective in diabetes patients in surgical processes. In this context, the study was designed to examine the effects of diabetes-based personalised discharge education given to surgical patients on satisfaction and diabetes empowerment.

DETAILED DESCRIPTION:
he population of the study consists of patients diagnosed with diabetes and undergoing surgery in the Surgical and Mixed service of Izzet Baysal Training and Research Hospital. The sample number of the experimental study, which was planned to be carried out between January 2025 and December 2026, was planned to include 100 patients with 0.05 error, 0.95 confidence interval and 0.85 power in the calculation made in the Gpower statistical programme based on previous studies. Considering that patients could leave the study for other reasons, it was decided to carry out the study by randomisation with 110 patients, which is 10% more.

Discharge Training Satisfaction Scale for Surgical Patients: It is a scale developed to measure the satisfaction of surgical patients with discharge training. It consists of 21 items in a five-point Likert structure and has been evaluated as a valid and reliable tool for measuring patient satisfaction. The scale covers factors such as discharge process, personal information, home care, infection monitoring and controls. The Cronbach α reliability coefficient was found to be 0.91, indicating that the scale is highly reliable Diabetes Empowerment Scale: It is a 5-point Likert-type scale consisting of 8 items. Turkish validity and reliability was carried out by Jahanpeyma et al. in 2020

ELIGIBILITY:
Inclusion Criteria:

* He's had an operation,
* Over 18 years old,
* Diagnosed with diabetes,
* Conscious patients returning to the clinic after surgery, not intubated

Exclusion Criteria:

* He's unconscious,
* Referral to intensive care,
* Patients who do not agree to participate in the study will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Discharge Training | through study completion, an average of 1 year
  It will be measured with the Discharge Training Satisfaction Scale Specific to Surgical Patients.
  Satisfaction will be measured with the 'Discharge Training Satisfaction Scale'. It consists of 21 items in a 5-point Likert scale. The scale does not contain negative items. The lowest score of 21 points and the highest score of 105 points can be obtained from the scale.
diabetes empowerment | through study completion, an average of 1 year
  The ability to manage the disease will be measured with the Diabetes Empowerment Scale.
  There are 28 items in Diabetes Empowerment Scale. Five-point Likert type (1:
  Strongly disagree, 5: Strongly agree), items 18,20,21,22,23,24,25,26 and 27 of this scale are under the sub-dimension of 'Self-awareness-managing psychological aspects of illness'; items 1,2,3,4,15,16,17 and 19 are under the sub-dimension of 'Ability to achieve goals'; items 5,6,7,8,9,10,11,12,13 and 14 are under the sub-dimension of 'Ability to set goals'.
  The minimum score of the scale is 28 and the maximum score is 140. A score between 28-65 points indicates a low level of resilience, 66-103 indicates a medium level, and 104-140 indicates a high level of resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data can be shared when requested by e-mail from the responsible author after the patient information is purified.